CLINICAL TRIAL: NCT04317027
Title: Physiological Examination of New Fighting Clothing During Exposure to Exercise Under Hot Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Dr. Sagi Arie Shpizer, Principal Investigator, Heller Institute of Medical Research, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHEBA-19-6652-SS-CTIL; 2017-2019-IDF (Registry Identifier: Israel Defense Forces (IDF))
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Clothing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): All subjects in this trial will receive the new fighting clothing while performing the study protocol
  Interventions: Device: New Fighting Clothing

INTERVENTIONS:
Device: New Fighting Clothing — VO2max test Clothing examination- 2-hour walk in 6 kph/4% elevation under 30 degrees Celsius and 60% relative humidity

SUMMARY:
The use of fighting clothing under extreme heat conditions during rest and exercise, compromises the body's ability to maintain temperature within the narrow physiological range needed for regular function, and might lead to heat injury. Beside working and fighting clothing, the fighters also wear vests used for protection and equipment carrying, which leads to substantial reduction in effective dissipation area from the central region of the body. This fact is most substantial during exercise which increases metabolic heat production rate and leads to heat accumulation and rise in body temperature. Therefore the development of new textile technologies to allow rapid cooling during intervals is of great importance.

This study is designed to physiologically examine new textile solutions, by evaluating the physiological stress induced during exercise under mild heat conditions.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Formerly fighters
* Healthy
* Without prior diseases including heart, vessel, respiratory and metabolic diseases or known use of medications
* experience in using fighting clothing
* VO2max > 50 ml/kg/min

Exclusion Criteria:

* Incapacity to fulfill inclusion criteria

Ages: 20 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Body temperature | During intervention period (2 hours test) only
  Using rectal thermometer
Heart rate | During intervention period (2 hours test) only
  Using heart rate watch

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Ha'Merkaz, Israel

IPD SHARING:
Plan to Share IPD: No